CLINICAL TRIAL: NCT05777044
Title: A Comparison of Hatha Yoga and Mediation on Mental Health Outcomes.
Brief Title: The Effect of Hatha Yoga on Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Danielle D Wadsworth, Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yoga RCT
Record Dates: First submitted 2023-03-09; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Depression; Anxiety; Mental Health Issue
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of three groups: waitlist control (usual routine), Hatha yoga (experimental group), and meditation (active comparative group).
Who Masked: Outcomes Assessor
Masking Description: Research personnel who administer heart rate variability and EEG were blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control- No Intervention/treatment (No Intervention): Participants in the control group will maintain their usual daily routine. The participants will complete the pre-test, 10 weeks of normal daily activities, and post-test. No changes to their daily schedule will be made by the researcher.
- Active Comparator- 10-week, 2x/week, 45-minute sessions of guided meditation (Active Comparator): The active comparator meditation group will complete a 10-week meditation yoga intervention (2x/week, 45 minutes per session). Each session will consist of yogic breathing, imagery, and meditation, specifically with a focus on each of the yogic limbs. The yogic limbs that will be incorporated during the meditation intervention are yamas, niyamas, pranayamas, and sense withdrawal/meditative techniques.
  Interventions: Behavioral: Yoga
- Experimental- 10-week, 2x/week, 45-minute Hatha yoga sessions (Experimental): The experimental hatha yoga group will complete a 10-week yoga intervention (2x/week, 45 minutes per session). Each session will consist of a centering, integration, awakening, vitality, equanimity, grounding, igniting, opening, release, and deep rest; all of which are specific hatha yoga practice sections. This group will complete the pre-test and post-test measures.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — Participation in Hatha Yoga twice a week for 45 minutes for 10 weeks. The total potential dose is 900 minutes over the course of the intervention.
  Arms: Active Comparator- 10-week, 2x/week, 45-minute sessions of guided meditation; Experimental- 10-week, 2x/week, 45-minute Hatha yoga sessions

SUMMARY:
The goal of this clinical trial is to determine the effects of a 10-week (2x a week; 45-minute per session) Hatha yoga intervention in adults ages 18-25 (n = 45) on mental health outcomes. The main questions it aims to answer are:

What is the effect of a hatha yoga intervention on depression and anxiety symptoms?

What is the effect of a hatha yoga intervention on electroencephalogram (EEG) alpha and theta band power?

What is the effect of hatha yoga intervention on heart rate variability?

Participants will be randomized to three groups: waitlist control (usual routine), Hatha yoga (experimental group), and meditation (active comparative group). Participants in the Hatha yoga experimental group will attend 10 weeks of twice-weekly 45-minute yoga sessions.

The active comparison meditation group will participate in 10 weeks of twice-weekly 45-minute meditation sessions. The control group will continue with their usual routine.

Researchers will compare changes in depression and anxiety symptoms, EEG alpha and theta band power, and heart rate variability between the three groups.

DETAILED DESCRIPTION:
There are knowledge gaps that need to be addressed in understanding the effects of yoga, specifically long-term interventions, on physiological markers, electroencephalography (EEG) and heart rate variability (HRV) and elevated mental health symptoms in young adults. The present study will address the knowledge gaps by evaluating the effect of a 10-week (2x a week; 45-minute per session) Hatha yoga intervention in adults ages 18-25 (n = 45). Participants will be truly randomized to three groups: waitlist control (usual routine), Hatha yoga (experimental group), and meditation (active comparative group). This design will allow the investigators to determine the effects of Hatha yoga on relevant outcome measures. Changes in depression symptoms (BDI), anxiety symptoms (BAI), EEG alpha and theta band power, heart rate variability indices (RMSSD, LF/HF) will be assessed. Compared to the control group, investigators hypothesize that both the Hatha yoga and meditation groups will exhibit an improvement in depression and anxiety symptoms, an increased alpha and theta band power at rest, and an increased RMSSD and decreased LF/HF at rest. Moreover, the investigators hypothesize that the Hatha yoga group will improve body composition, flexibility, muscular endurance and strength, and cardiovascular recovery more than the meditation group.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-35
* Medically healthy to participate in physical activity as determined by the Physical Activity Reading Questionnaire (PAR-Q)
* Concerned about or experiencing heightened anxiety, depression, and/or stress symptoms

Exclusion Criteria:

* Those with diagnosed with an intellectual or developmental disability, currently diagnosed with a concussion, physically unhealthy to participate in physical activity
* Anyone currently taking beta-blockers

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
EEG | 10 weeks
  Frontal (F7/F8) and Temporoparietal (TP9/TP10) Alpha and Theta EEG power. 5-minute recording at rest; measured using the MUSE-2 system and Mind Monitor application.
Heart rate variability | 10 weeks
  Root mean square of successive differences (RMSSD) and low-frequency/high-frequency ratio (LF/HF) indices of heart rate variability (HRV), 5-minute recording at rest; measured using the Polar H8/H9 HR monitors and HRVLogger application.
Depression | 10 weeks
  Beck's Depression Inventory (BDI) scores as measured by the Beck's Depression Inventory
Anxiety | 10 weeks
  Beck's Anxiety Inventory (BAI) scores as measured by the Beck's Anxiety Inventory

SECONDARY OUTCOMES:
Blood Pressure | 10 weeks
  Resting blood pressure will be assessed with a automatic blood pressure cuff.
Body Fat Percentage | 10 weeks
  • Body Composition as measured by changes in body fat percentage (ratio of lean mass to fat mass)
Flexbility | 10 weeks
  Changes in shoulder and hamstring flexibility assessed with the Fitnessgram.
Muscular Endurance | 10 weeks
  Changes in push-up fitnessgram tests
Aerobic capacity | 10 weeks
  3-minute YMCA step-test which will be an index of aerobic capacity

CONTACTS AND LOCATIONS:
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.